CLINICAL TRIAL: NCT00603941
Title: A Phase 1/2 Study of CS7017, an Oral PPARγ Agonist, in Combination With Paclitaxel in Subjects With Advanced Anaplastic Thyroid Cancer
Brief Title: A Phase 1/2 Study of CS7017, an Oral PPARγ Agonist, in Combination With Paclitaxel
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Due to low enrollment, no participant had a dose limiting toxicity, therefore a maximum tolerated dose could not be established
Sponsor: Daiichi Sankyo (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CS7017-A-U103
Record Dates: First submitted 2008-01-15; First posted 2008-01-29 (Estimated); Results first posted 2020-09-16 (Actual); Last update posted 2020-09-16 (Actual); Status verified 2020-08

CONDITIONS: Anaplastic Thyroid Cancer
Keywords: Anaplastic Thyroid Cancer; Neoplasm; Tumor; Anti-neoplastic Agent; First-line treatment of advanced Anaplastic thyroid cancer
MeSH Terms: conditions — Thyroid Carcinoma, Anaplastic; Neoplasms | interventions — efatutazone; Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Cohort 1; 0.15 mg CS-7017 (Experimental): Participants who received 0.15 mg twice daily (BID) oral CS-7017 and 135 [Dose Level 1a] or 175 [Dose Level 1b] mg/m^2 intravenous (IV) paclitaxel once every 3 weeks.
  Interventions: Drug: CS-7017; Drug: Paclitaxel
- Cohort 2; 0.30 mg CS-7017 (Experimental): Participants who received 0.30 mg twice daily (BID) oral CS-7017 and 175 mg/m^2 IV paclitaxel once every 3 weeks.
  Interventions: Drug: CS-7017; Drug: Paclitaxel
- Cohort 3; 0.50 mg CS-7017 (Experimental): Participants who received 0.50 mg twice daily (BID) oral CS-7017 and 175 mg/m^2 IV paclitaxel once every 3 weeks.
  Interventions: Drug: CS-7017; Drug: Paclitaxel

INTERVENTIONS:
Drug: CS-7017 — At Phase 1, CS-7017 will be tested in combination with paclitaxel at the following dosage levels: 0.15, 0.30, or 0.50 mg BID. At Phase 2, CS-7017 will be administered at the recommended phase 2 dose (RP2D).
Drug: Paclitaxel — Commercially available paclitaxel will be administrated as IV infusion over 3 hours once every 3 weeks.

SUMMARY:
The Phase I/II study will be conducted as an open label, multiple center study of CS-7017, an experimental drug and paclitaxel chemotherapy in subjects with advanced anaplastic thyroid cancer. Biopsies will be obtained from patients with accessible tumor at baseline, two-weeks after the first CS-7017 dosage (prior to the start of combination therapy) and at the end of the first study cycle (week 3 of combination therapy), in order to evaluate the effects of the study drug alone and in combination with the chemotherapy agent on the tumor. Treatment will continue until disease progression or the development of intolerable toxicities.

ELIGIBILITY:
During the Phase 1 and Phase 2 portions of the study, participant eligibility criteria are identical except for prior treatment for anaplastic thyroid cancer (ATC). During Phase 1, eligible participants may have received prior chemotherapy while during Phase 2, eligible participants must be chemotherapy naïve.

Inclusion Criteria:

* Histologically or cytologically diagnosed, advanced ATC
* Measurable lesion(s)
* Lesion(s) (primary or metastatic) with viable tumor tissue accessible for repeated biopsy
* Age equal to or older than 18 years
* Eastern Cooperative Oncology Group (ECOG) performance status less than or equal to 2
* Adequate organ and bone marrow function
* Agreement to use effective contraception while on treatment and for equal to or greater than 3 months after end of treatment
* Pregnant or breastfeeding

Exclusion Criteria:

* Medical history of diabetes mellitus requiring treatment with insulin or oral agents; no pleural or pericardial effusion or clinically significant pulmonary or cardiovascular disease.
* Clinically active brain metastasis, uncontrolled seizure disorder, spinal cord compression, or carcinomatous meningitis
* Clinically significant active infection requiring antibiotic or antiretroviral therapy
* Concomitant use of other thiazolidinediones (TZDs)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2008-01; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Director Clinical Development, Study Director — Daiichi Sankyo
Locations (10):
- United States (10):
  - Univ of Colorado Cancer Center, Aurora, Colorado
  - Mayo Clinic, Jacksonville, Florida
  - Massachusetts General Hospital, Boston, Massachusetts
  - Mayo Clinic, Rochester, Minnesota
  - Washington University, Siteman Cancer Center, St Louis, Missouri
  - Ohio State Univ, Columbus, Ohio
  - Oregon Health Science Univ, Portland, Oregon
  - University of Pennsylvania Maloney Hospital, Philadelphia, Pennsylvania
  - Vanderbilt Ingram Cancer Center, Nashville, Tennessee
  - Eastern Virginia Medical School, Norfolk, Virginia

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) and applicable supporting clinical trial documents may be available upon request at https://vivli.org/. In cases where clinical trial data and supporting documents are provided pursuant to our company policies and procedures, Daiichi Sankyo will continue to protect the privacy of our clinical trial participants. Details on data sharing criteria and the procedure for requesting access can be found at this web address: https://vivli.org/ourmember/daiichi-sankyo/
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Studies for which the medicine and indication have received European Union (EU) and United States (US), and/or Japan (JP) marketing approval on or after 01 January 2014 or by the US or EU or JP Health Authorities when regulatory submissions in all regions are not planned and after the primary study results have been accepted for publication.
Access Criteria: Formal request from qualified scientific and medical researchers on IPD and clinical study documents from clinical trials supporting products submitted and licensed in the United States, the European Union and/or Japan from 01 January 2014 and beyond for the purpose of conducting legitimate research. This must be consistent with the principle of safeguarding study participants' privacy and consistent with provision of informed consent.
URL: https://vivli.org/ourmember/daiichi-sankyo/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 19 participants who met all inclusion and no exclusion criteria were enrolled in the study; 15 received treatment.
  Due to low enrollment, no participant had a dose limiting toxicity, therefore a maximum tolerated dose required for the recommendation of Phase 2 dose could not be established. Therefore, the study was halted prematurely.
Pre-assignment Details: Sequential cohorts per dose level were treated with CS-7017 and paclitaxel in accordance with prospectively defined dose levels, dose escalation rules, and definitions of treatment-related dose-limiting toxicity (DLT).
Groups:
- Cohort 1; 0.15 mg CS-7017: Participants who received 0.15 mg twice daily (BID) oral CS-7017 and 135 [Dose Level 1a] or 175 [Dose Level 1b] mg/m^2 IV paclitaxel once every 3 weeks.
Period: Overall Study
Arm/Group | Cohort 1; 0.15 mg CS-7017 | Cohort 2; 0.30 mg CS-7017 | Cohort 3; 0.50 mg CS-7017
Started | 7 | 10 | 2
Completed | 0 | 0 | 0
Not Completed | 7 | 10 | 2
Not completed — Disease progression | 6 | 7 | 1
Not completed — Adverse Event | 1 | 0 | 1
Not completed — Physician Decision | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 2 | 0

BASELINE CHARACTERISTICS:
Population: Baseline characteristics are reported for the Safety Analysis Set.
Groups:
- Cohort 1; 0.15 mg CS-7017: Participants who received 0.15 mg BID oral CS-7017 and 135 [Dose Level 1a] or 175 [Dose Level 1b] mg/m^2 IV paclitaxel once every 3 weeks.
- Cohort 2; 0.30 mg CS-7017: Participants who received 0.30 mg BID oral CS-7017 and 175 mg/m^2 IV paclitaxel once every 3 weeks.
- Cohort 3; 0.50 mg CS-7017: Participants who received 0.50 mg BID oral CS-7017 and 175 mg/m^2 IV paclitaxel once every 3 weeks.
- Total: Total of all reporting groups
Arm/Group | Cohort 1; 0.15 mg CS-7017 | Cohort 2; 0.30 mg CS-7017 | Cohort 3; 0.50 mg CS-7017 | Total
Number analyzed (Participants) | 7 | 6 | 2 | 15
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 5 | 4 | 0 | 9
  >=65 years | 2 | 2 | 2 | 6
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.6 (12.79) | 59.8 (8.75) | 73.5 (0.71) | 61.1 (11.11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 4 | 2 | 10
  Male | 3 | 2 | 0 | 5
Region of Enrollment [Number; unit: participants]
  United States | 7 | 6 | 2 | 15

OUTCOME MEASURES:

1. Primary Outcome: Overall Progression-free Survival in Participants After a Dosage of CS-7017 Administered Twice Daily in Combination With Paclitaxel Administered Once Every 3 Weeks to Participants With Advanced Anaplastic Thyroid Cancer (ATC)
Description: Progression-free survival (PFS) was defined as the time from enrollment to the date of the first objective documentation of disease progression or death resulting from any cause, whichever comes first. Progression was defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) as at least a 20% increase in the sum of diameters of target lesions.
Time Frame: From baseline up to disease progression or death, up to approximately 2 years postdose
Population: PFS was assessed in the Efficacy Analysis Set. Since the study halted prematurely due to low enrollment and failed to establish a recommendation for a Phase 2 dose, it was not feasible to analyze the primary outcomes per arm. The arms were combined post hoc based on these circumstances and primary efficacy outcomes were assessed in all patients.
Measure: Median (95% Confidence Interval); unit: days
Groups:
- All Patients: All patients who received any dose of CS-7017 combined with paclitaxel chemotherapy.
Arm/Group | All Patients
Number analyzed (Participants) | 15
days | 55.5 [29.0 to 71.0]

2. Primary Outcome: Overall Survival in Participants After a Dosage of CS-7017 Administered Twice Daily in Combination With Paclitaxel Administered Once Every 3 Weeks to Participants With Advanced Anaplastic Thyroid Cancer (ATC)
Description: Overall survival (OS) was defined as the time from the date enrollment to the date of death.
Time Frame: From baseline up to date of death, up to approximately 2 years postdose
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | All Patients
Number analyzed (Participants) | 15
days | 130.0 [99.0 to 142.0]

3. Primary Outcome: Best Overall Response in Participants After a Dosage of CS-7017 Administered Twice Daily in Combination With Paclitaxel Administered Once Every 3 Weeks to Participants With Advanced Anaplastic Thyroid Cancer (ATC)
Description: The best overall response was the best response (in the order of confirmed complete response [CR], confirmed partial response [PR], stable disease [SD], and progressive disease [PD]) among all overall responses recorded from the start of treatment until the subject withdraws from the study. If there is no tumor assessment after the date of enrollment, the best overall response is classified as Unknown.
Time Frame: From baseline up to disease progression or the development of unacceptable toxicity, up to approximately 2 years postdose
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | All Patients
Number analyzed (Participants) | 15
Participants
  Confirmed complete response (CR) | 0
  Confirmed partial response (PR) | 1
  Objective response (confirmed CR + PR) | 1
  Stable disease | 8
  Progressive disease | 4
  Unknown | 2

4. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events, Summarized by Worst CTCAE Grade (≥3) and Preferred Term After Administration of CS-7017 Combined With Paclitaxel Administered to Participants With Advanced Anaplastic Thyroid Cancer (ATC)
Description: Treatment-emergent adverse events (TEAEs) are defined as adverse events that started or worsened after the first dose of any study drug (after Day 1 or first day of CS-7017 monotherapy) but adverse events occurring more than 30 days after the last dose are not considered TEAEs unless also considered to be related (possibly, probably, or definitely) to study drug.
Time Frame: From baseline up to 30 days after last dose, up to approximately 2 years
Population: TEAEs were assessed in the Safety Analysis Set.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1; 0.15 mg CS-7017 | Cohort 2; 0.30 mg CS-7017 | Cohort 3; 0.50 mg CS-7017
Number analyzed (Participants) | 7 | 6 | 2
Participants
  Any Severe TEAE of Grade ≥3 | 3 | 5 | 2
  Anaemia | 0 | 1 | 0
  Dysphagia | 1 | 0 | 0
  Disease progression | 2 | 0 | 0
  Anaphylatic reaction | 0 | 0 | 1
  Pneumonia | 0 | 1 | 0
  Septic shock | 1 | 0 | 0
  Neutrophil count decreased | 0 | 1 | 0
  Loss of consciousness | 0 | 0 | 1
  Dyspnoea | 0 | 1 | 0

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse event data were collected from baseline up to 30 days after last dose, up to approximately 2 years.
Description: Adverse events (AEs) were defined as any untoward, unfavorable, unintended medical occurrence in a participant administered a pharmaceutical product and which does not necessarily have to have a causal relationship with this treatment. All-cause mortality includes all deaths that occurred during the study and within 30 days after the last dose of study drug.
Arm/Group | Cohort 1; 0.15 mg CS-7017 | Cohort 2; 0.30 mg CS-7017 | Cohort 3; 0.50 mg CS-7017
All-Cause Mortality (participants affected / at risk) | 6/7 | 6/6 | 0/2
Serious Adverse Events (participants affected / at risk) | 3/7 | 3/6 | 2/2
Other Adverse Events (participants affected / at risk) | 6/7 | 6/6 | 2/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1; 0.15 mg CS-7017 (N=7) | Cohort 2; 0.30 mg CS-7017 (N=6) | Cohort 3; 0.50 mg CS-7017 (N=2)
Confusional state (Psychiatric disorders) | 1 | 0 | 0
Septic shock (Infections and infestations) | 1 | 0 | 0
Disease progression (General disorders) | 2 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 1 | 0 | 0
Clostridial infection (Infections and infestations) | 0 | 1 | 0
Pneumonia (Infections and infestations) | 0 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0
Loss of consciousness (Nervous system disorders) | 0 | 0 | 1
Anaphylatic reaction (Immune system disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1; 0.15 mg CS-7017 (N=7) | Cohort 2; 0.30 mg CS-7017 (N=6) | Cohort 3; 0.50 mg CS-7017 (N=2)
Anaemia (Blood and lymphatic system disorders) | 2 | 1 | 0
Leukopenia (Blood and lymphatic system disorders) | 2 | 0 | 0
Lymphopenia (Blood and lymphatic system disorders) | 1 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 1 | 0
Constipation (Gastrointestinal disorders) | 2 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 1 | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 3 | 0
Disease progression (General disorders) | 2 | 0 | 0
Face oedema (General disorders) | 2 | 0 | 0
Fatigue (General disorders) | 2 | 4 | 2
Feeling cold (General disorders) | 1 | 0 | 0
Oedema peripheral (General disorders) | 1 | 3 | 0
Pitting oedema (General disorders) | 1 | 0 | 0
Pneumonia (Infections and infestations) | 1 | 1 | 0
Septic shock (Infections and infestations) | 1 | 0 | 0
Haemoglobin decreased (Investigations) | 1 | 2 | 0
International normalised ratio increased (Investigations) | 1 | 0 | 0
Prothrombin time prolonged (Investigations) | 1 | 0 | 0
Weight decreased (Investigations) | 1 | 1 | 0
Weight increased (Investigations) | 1 | 3 | 0
Hyperlipidaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 1 | 1 | 0
Hypovolaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 1 | 0
Groin pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Anxiety (Psychiatric disorders) | 1 | 1 | 0
Confusional state (Psychiatric disorders) | 1 | 0 | 0
Insomnia (Psychiatric disorders) | 1 | 2 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Throat tightness (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 3 | 2 | 0
Erythema (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Pain of skin (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 1 | 0
Localised oedema (General disorders) | 0 | 1 | 0
Pyrexia (General disorders) | 0 | 1 | 0
Cellulitis (Infections and infestations) | 0 | 1 | 0
Clostridial infection (Infections and infestations) | 0 | 1 | 0
Rhinitis (Infections and infestations) | 0 | 1 | 0
Blood creatinine increased (Investigations) | 0 | 1 | 0
Blood urea increased (Investigations) | 0 | 1 | 0
Neutrophil count decreased (Investigations) | 0 | 1 | 0
Platelet count decreased (Investigations) | 0 | 1 | 0
Anorexia (Metabolism and nutrition disorders) | 0 | 1 | 0
Fluid retention (Metabolism and nutrition disorders) | 0 | 1 | 0
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Joint stiffness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Dizziness (Nervous system disorders) | 0 | 1 | 1
Headache (Nervous system disorders) | 0 | 1 | 1
Hypoaesthesia (Nervous system disorders) | 0 | 1 | 0
Neuropathy peripheral (Nervous system disorders) | 0 | 2 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 1 | 0
Depression (Psychiatric disorders) | 0 | 2 | 0
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 4 | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Swelling face (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Hypotension (Vascular disorders) | 0 | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 1
Anaphylactic reaction (Immune system disorders) | 0 | 0 | 1
Loss of consciousness (Nervous system disorders) | 0 | 0 | 1
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1

LIMITATIONS AND CAVEATS:
The study was halted prematurely due to low enrollment and failure to establish recommendation of Phase 2 dose. Analysis for the primary efficacy outcomes were also combined for the study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No